CLINICAL TRIAL: NCT07245745
Title: Prospective Clinical Study Comparing Patient-reported Outcomes Measurements (PROMS) After Adaptive or Conventional Radiotherapy in Prostate Cancer
Brief Title: Prospective Clinical Study Comparing PROMS After Adaptive or Conventional Radiotherapy in Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/27MAI/209
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm H-RT (Active Comparator): Treatment planned and delivered on the Halcyon machine with non-adaptive conventional radiotherapy.
  Interventions: Radiation: Radiotherapy
- Arm E-ART (Active Comparator): Treatment planned and delivered on the Ethos machine with adaptive radiotherapy.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Prostate cancer patients will be treated radiotherapy.

SUMMARY:
This prospective clinical study compares patient-reported outcome measures (PROMs) after adaptive or conventional radiotherapy in prostate cancer. Adaptive radiotherapy (ART) aims to reduce uncertainties related to daily anatomical variations, thereby improving treatment accuracy while decreasing gastrointestinal (GI) and genitourinary (GU) toxicity. This study, conducted at Cliniques universitaires Saint-Luc (Brussels and Ottignies sites), analyzes and compares toxicities in patients treated with ART on Ethos and those treated with conventional radiotherapy on Halcyon.

The primary objective of the study is to demonstrate that ART reduces gastrointestinal, urinary, and general side effects induced by radiotherapy. Additionally, the secondary objectives include assessing the duration of these effects, correlating them with dosimetric data, analyzing the management of toxicities through the Noona e-health application, as well as evaluating the use of this application by both patients and healthcare providers.

The study includes men aged 18 years or older with prostate cancer undergoing curative-intent treatment, with an ECOG performance status of 0 to 1, and able to use the Noona application. Patients with a history of rectal or bladder treatment, or those who have already received pelvic radiotherapy, are excluded. Two groups are compared: patients treated with conventional radiotherapy on Halcyon (Ottignies site) and those treated with adaptive radiotherapy on Ethos (Brussels site).

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer referred for curative-intent radiotherapy
* Male patients ≥ 18 years old
* ECOG performance status 0-1
* Patients willing to use an e-health application
* Patients capable of using an e-health application
* Proficient in French, English, or Dutch
* No prior history of treatment for rectal or bladder cancer
* No prior history of pelvic radiotherapy

Exclusion Criteria:

* Cognitive impairment
* ECOG ≥ 2
* History of treatment for rectal or bladder cancer
* History of pelvic radiotherapy
* No access to the Noona application on a smartphone or computer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Demonstration that adaptive radiotherapy in prostate cancer helps reduce radiotherapy-induced side effects (digestive, urinary, and general toxicity) using PROMS questionnaires. | 3 years
  In this clinical study, we aim to demonstrate that adaptive radiotherapy (ART) in prostate cancer can reduce radiotherapy-induced side effects (digestive, urinary, and general toxicity). Daily adaptation of treatment plans not only ensures better target coverage but also accounts for daily variations in the position or deformation of organs at risk (OARs). Consequently, ART could reduce the occurrence of genitourinary (GU) and gastrointestinal (GI) side effects, either early (during or shortly after treatment) or at later stages (up to one year after completion of treatment). Three questionnaires will be used: the Expanded Prostate Cancer Index Composite-26 (EPIC-26), the EuroQol 5 Dimensions (EQ-5D) and the International Prostate Symptom Score (IPSS).

SECONDARY OUTCOMES:
Evaluation of the time to recovery from treatment-related adverse effects using PROMS questionnaires. | 3 years
  This study will collect PROMs and clinical data to assess whether the duration of adverse effects before recovery differs between the two radiotherapy approaches (adaptive versus conventional).
Correlation of the duration of adverse effects collected with PROMS questionnaire with the dosimetric data. | 3 years
  The duration of adverse effects before recovery may also be correlated with dosimetric analyses. Indeed, ART could allow better dose coverage of the target volumes while reducing the dose delivered to the OARs. The Ethos system enables monitoring of the accumulated dose to both targets and OARs, thereby allowing complementary dosimetric analyses.
Evaluation of the management of treatment-related toxicity using the e-health application using a PREM questionnaire at the end of the study. | 3 years
  Since patients will complete PROMs questionnaires through an e-health application, this will allow a qualitative analysis of the application. Specific questions will be asked to patients regarding their use of the application.
Number of participants and medical staff satisfied by the ease of use of an e-health application during radiotherapy using a questionnaire. | 3 years
  This study could thus highlight a novel approach to managing patient toxicity and assess whether it could improve overall treatment management.

CONTACTS AND LOCATIONS:
Overall Officials: Heylen Sofie, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Background] de Crevoisier R, Tucker SL, Dong L, Mohan R, Cheung R, Cox JD, Kuban DA. Increased risk of biochemical and local failure in patients with distended rectum on the planning CT for prostate cancer radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):965-73. doi: 10.1016/j.ijrobp.2004.11.032. PMID 15989996
- [Background] Heemsbergen WD, Hoogeman MS, Witte MG, Peeters ST, Incrocci L, Lebesque JV. Increased risk of biochemical and clinical failure for prostate patients with a large rectum at radiotherapy planning: results from the Dutch trial of 68 GY versus 78 Gy. Int J Radiat Oncol Biol Phys. 2007 Apr 1;67(5):1418-24. doi: 10.1016/j.ijrobp.2006.11.014. Epub 2007 Jan 22. PMID 17241751
- [Background] Yan D, Vicini F, Wong J, Martinez A. Adaptive radiation therapy. Phys Med Biol. 1997 Jan;42(1):123-32. doi: 10.1088/0031-9155/42/1/008. PMID 9015813
- [Background] Posiewnik M, Piotrowski T. A review of cone-beam CT applications for adaptive radiotherapy of prostate cancer. Phys Med. 2019 Mar;59:13-21. doi: 10.1016/j.ejmp.2019.02.014. Epub 2019 Feb 22. PMID 30928061
- [Background] Byrne M, Archibald-Heeren B, Hu Y, Teh A, Beserminji R, Cai E, Liu G, Yates A, Rijken J, Collett N, Aland T. Varian ethos online adaptive radiotherapy for prostate cancer: Early results of contouring accuracy, treatment plan quality, and treatment time. J Appl Clin Med Phys. 2022 Jan;23(1):e13479. doi: 10.1002/acm2.13479. Epub 2021 Nov 29. PMID 34846098
- [Background] Thornqvist S, Hysing LB, Tuomikoski L, Vestergaard A, Tanderup K, Muren LP, Heijmen BJ. Adaptive radiotherapy strategies for pelvic tumors - a systematic review of clinical implementations. Acta Oncol. 2016 Aug;55(8):943-58. doi: 10.3109/0284186X.2016.1156738. Epub 2016 Apr 8. PMID 27055486
- [Background] Christiansen RL, Dysager L, Hansen CR, Jensen HR, Schytte T, Nyborg CJ, Bertelsen AS, Agergaard SN, Mahmood F, Hansen S, Hansen O, Brink C, Bernchou U. Online adaptive radiotherapy potentially reduces toxicity for high-risk prostate cancer treatment. Radiother Oncol. 2022 Feb;167:165-171. doi: 10.1016/j.radonc.2021.12.013. Epub 2021 Dec 16. PMID 34923034
- [Background] Brunelli C, Zito E, Alfieri S, Borreani C, Roli A, Caraceni A, Apolone G. Knowledge, use and attitudes of healthcare professionals towards patient-reported outcome measures (PROMs) at a comprehensive cancer center. BMC Cancer. 2022 Feb 10;22(1):161. doi: 10.1186/s12885-022-09269-x. PMID 35144569